CLINICAL TRIAL: NCT00843518
Title: Assessment of LY451395 for Neuropsychiatric Symptoms of Aggression and Agitation in Alzheimer's Disease
Brief Title: Treatment for Aggression and Agitation in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12541; H6N-MC-LEAQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Alzheimer's Disease
Keywords: Agitation and Aggression
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Aggression | interventions — N-((2-(4'-(2-(methylsulfonyl)amino)ethyl)(1,1'-biphenyl)-4-yl)propyl)-2-propanesulfonamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY451395 (Experimental): 3 milligram (mg) LY451395 orally twice daily for 12 weeks; may have been reduced to 1 mg if participant was unable to tolerate
  Interventions: Drug: LY451395
- Placebo (Placebo Comparator): Placebo orally twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY451395 — 3 mg LY451395 orally twice daily for 12 weeks; may have been reduced to 1 mg if participant was unable to tolerate
  Other Names: mibampator
  Arms: LY451395
Drug: Placebo — Placebo orally twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether this drug can help symptoms of aggression and agitation in participants with Alzheimer's disease.

DETAILED DESCRIPTION:
The primary purpose of this study is to help answer the following research questions:

* Whether this drug can help symptoms of aggression and agitation in participants with Alzheimer's Disease.
* The safety of this drug and any side effects that might be associated with it.
* How this drug compares to placebo.

During the 12-week period of this study, the participant will have an equal chance of receiving 1 of the 2 treatment groups: active drug or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling participants with a diagnosis of probable Alzheimer's disease (AD) based on disease criteria from the National Institute of Neurological and Communicative Disorders and Stroke (NINCDS) and the Alzheimer's Association. Mini Mental State Examination (MMSE) score from 6 to 26 inclusive; Neuropsychiatric Inventory-10 (NPI-10) total score greater than or equal to 10.
* Are men or women at least 60 years old.
* Weight greater than or equal to 45 kilograms (kg).
* Have clinically significant and persistent verbal or physical agitation and/or verbal or physical aggression behaviors that are disruptive to daily functioning or potentially harmful and occurred at least 3 days per week over the past 4 weeks prior to study entry.
* Understand English.
* Have a reliable and actively involved caregiver who must be able to communicate in English and be willing to comply with protocol requirements.

Exclusion Criteria:

* Meet DSM-IV-TR or Delirium Rating Scale-Revised-98 criteria for delirium.
* Does not score ≤4 on the Modified Hachinski Ischemia Scale for vascular dementia.
* Have a magnetic resonance imaging (MRI) or computer tomography (CT) scan on file since the onset of symptoms of AD and performed within the past 24 months that is inconsistent with a diagnosis of AD.
* Have a current, required use, or expected use of psychoactive drugs or other medications not allowed in this trial.
* Have currently active significant medical, neurological, or psychiatric problems that are not allowed in this trial or other brain disorders.
* Have received acetylcholinesterase inhibitor (AChEIs) or memantine for less than 4 months, or have less than 2 months of stable therapy on these treatments by Visit 2.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877.CTLilly (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM-5PM Easter time (UTC/GMT-5 hours, EST, Study Director — Eli Lilly and Company
Locations (17):
- United States (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Costa Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamden, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Easton, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flowood, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hickory, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norristown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bennington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waukesha, Wisconsin

REFERENCES:
- [Derived] Trzepacz PT, Cummings J, Konechnik T, Forrester TD, Chang C, Dennehy EB, Willis BA, Shuler C, Tabas LB, Lyketsos C. Mibampator (LY451395) randomized clinical trial for agitation/aggression in Alzheimer's disease. Int Psychogeriatr. 2013 May;25(5):707-19. doi: 10.1017/S1041610212002141. Epub 2012 Dec 21. PMID 23257314

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period 1 lasted 3 to 28 days and included screening tests and procedures (N=205). Study Period 2 was a 12-week, randomized, double-blind treatment period with clinic visits at 3-week intervals and intervening weekly telephone assessments with caregivers (N=132). Study Period 3 was a 1-week, single-blind washout period (N=91).
Groups:
- LY451395: 3 milligram (mg) LY451395 (mibampator) orally twice daily for 12 weeks; may have been reduced to 1 mg if participant was unable to tolerate
Period: Period 2 (Double-blind Treatment)
Arm/Group | LY451395 | Placebo
Started | 63 | 69
Completed | 43 | 49
Not Completed | 20 | 20
Not completed — Adverse Event | 5 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 2 | 5
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Caregiver decision | 7 | 7
Period: Period 3 (Single-blind Washout)
Arm/Group | LY451395 | Placebo
Started | 42 (1 LY451395 participant completed double-blind treatment, but did not enter washout period.) | 49
Completed | 42 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY451395 | Placebo | Total
Number analyzed (Participants) | 63 | 69 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.21 (8.246) | 77.66 (7.574) | 77.44 (7.874)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 36 | 67
  Male | 32 | 33 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 61 | 69 | 130
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 53 | 62 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 63 | 69 | 132
Mini Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — MMSE assessed cognitive function in elderly participants. The scale ranged from 0 to 30, with higher scores indicating higher cognitive function.
  units on a scale | 16.0 (6.06) | 18.0 (5.26) | 17.0 (5.72)
4-Item version of Neuropsychiatric Inventory (NPI-4) of Agitation and Aggression (A/A) [Mean (Standard Deviation); unit: units on a scale] — NPI assessed noncognitive psychopathology in participants with Alzheimer's dementia. A 4-item subscale of the standard 12-item NPI measured the neuropsychiatric symptoms of A/A, with items consisting of agitation/aggression, aberrant motor behavior, irritability/emotional lability, and disinhibition. Scores for each subscale (frequency x severity) were calculated to obtain each item score. The total subscale score ranged from 0 to 48, with higher scores indicating more frequent and/or severe A/A symptoms. If a symptom was not present at all then a zero would be imputed for that item.
  units on a scale | 18.8 (8.72) | 18.1 (8.19) | 18.4 (8.42)
10-Item version of Neuropsychiatric Inventory (NPI-10) [Mean (Standard Deviation); unit: units on a scale] — NPI assessed noncognitive psychopathology in participants with Alzheimer's dementia. A 10-item scale of the standard 12-item NPI measured neuropsychiatric symptoms minus appetite and sleep disturbance. Scores for each subscale (frequency × severity) were calculated to obtain the item score. The total subscale score ranged from 0 to 120, with higher scores indicating more frequent and/or severe A/A symptoms. If a symptom was not present at all, the site would not enter anything for frequency or severity, and a zero would be imputed for that item.
  units on a scale | 31.9 (16.67) | 29.7 (13.22) | 30.7 (14.95)
Neuropsychiatric Inventory (NPI) Depression Domain [Mean (Standard Deviation); unit: units on a scale] — NPI Depression domain was an item of the standard 12-item NPI that measured depression in participants with Alzheimer's dementia. Scores for each subscale (frequency x severity) were calculated to obtain the item score, which ranged from 0 to 12, with higher scores indicating more frequent and/or severe neuropsychiatric symptoms.
  units on a scale | 2.2 (3.10) | 1.8 (2.33) | 2.0 (2.73)
Neuropsychiatric Inventory (NPI) Psychosis Subscale [Mean (Standard Deviation); unit: units on a scale] — The NPI Psychosis subscale score was the sum of the delusions and hallucinations items of the standard 12-item NPI that measured psychosis symptoms in participants with Alzheimer's dementia. Scores for each subscale (frequency x severity) were calculated for each item score and ranged from 0 to 24 with higher scores indicating more frequent and/or severe neuropsychiatric symptoms.
  units on a scale | 3.2 (5.24) | 2.4 (3.92) | 2.8 (4.60)
Cohen-Mansfield Agitation Inventory-Community (CMAI-C) Version [Mean (Standard Deviation); unit: units on a scale] — CMAI-C is the Cohen-Mansfield Agitation Inventory - Community Version, and it contained 36 questions. The first 35 items were rated from 1 (never) to 7 (several times per hour) and the last item asked if there was any other inappropriate behavior, with a free text field to specify the behavior. The total score ranged from 7 to 245 (7 x 35), with higher scores reflecting more severe agitation.
  units on a scale | 73.6 (22.55) | 64.7 (17.58) | 68.9 (20.52)
Cornell Scale for Depression in Dementia (CSDD) [Mean (Standard Deviation); unit: units on a scale] — CSDD was a 19-item, clinician-rated scale designed to measure the presence and severity of depressive symptoms in dementia participants. Symptoms were rated as absent, mild/intermittent, or severe. Scores ranged from 0 to 38; scores of 8 or more suggested clinical depression.
  units on a scale | 8.4 (5.40) | 8.0 (4.63) | 8.2 (4.99)
Total T-Score in the Frontal System Behaviors (FrSBe) Scale [Mean (Standard Deviation); unit: units on a scale] — FrSBe was a 46-item, caregiver-rated scale that assessed behaviors associated with damage to the frontal lobes and frontal systems of the brain, including executive function, disinhibition, and apathy. Raw scores were normalized to T-scores based on gender, education, and age. Higher T scores represent a worse outcome. A score of 50 reflects a normative sample, and T scores at or above 65 are considered clinically significant.
  units on a scale | 92.4 (22.50) | 89.1 (18.50) | 90.7 (22.11)
Clinical Global Impression-Severity-Agitation/Aggressive (CGI-S-A/A) [Mean (Standard Deviation); unit: units on a scale] — CGI-S-A/A was a 7-point, single-item rating scale for overall severity of symptoms based on the investigator's general clinical experience with a similar participant population. This Likert scale ranged from 0 (normal) to 7 (most severely ill).
  units on a scale | 4.1 (0.68) | 4.1 (0.69) | 4.1 (0.68)
Clinical Global Impression-Severity-Global Functioning (CGI-S-GF) [Mean (Standard Deviation); unit: units on a scale] — CGI-S-GF was a 7-point, single-item rating scale for overall functioning based on the investigator's general clinical experience with a similar participant population. This Likert scale ranged from 0 (normal) to 7 (most severely ill).
  units on a scale | 4.1 (0.88) | 4.0 (0.78) | 4.1 (0.82)
14-Item Alzheimer's Disease Assessment Scale, Cognitive Subscale (ADAS-Cog14) [Mean (Standard Deviation); unit: units on a scale] — ADAS-Cog14, a 14-item rating scale, measured the severity of cognitive dysfunction in persons with Alzheimer's disease (AD). Scores ranged from 0 to 90, with a higher score indicating worse cognitive functioning.
  units on a scale | 43.3 (20.42) | 40.0 (18.07) | 41.6 (19.22)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the 4-Item Agitation/Aggression Subscale of the Neuropsychiatric Inventory (NPI-4 A/A) at Week 12
Description: NPI assessed noncognitive psychopathology in participants with Alzheimer's dementia. A 4-item subscale of the standard 12-item NPI measured the neuropsychiatric symptoms of A/A, with items consisting of agitation/aggression, aberrant motor behavior, irritability/emotional lability, and disinhibition. Scores for each subscale (frequency x severity) were calculated to obtain each item score. The total subscale score ranged from 0 to 48, with higher scores indicating more frequent and/or severe A/A symptoms. If a symptom was not present at all, the site would not enter anything for frequency or severity, and a zero would be imputed for that item. Least Squares (LS) Mean value was adjusted for NPI strata, treatment, pooled site, visit, treatment-by-visit, baseline NPI-4 A/A, and baseline-by-visit interaction.
Time Frame: Baseline, Week 12
Population: The analysis population included all randomized participants and was a modified intent-to-treat (ITT) population defined as having both a baseline and at least 1 post-baseline measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY451395 | Placebo
Number analyzed (Participants) | 43 | 50
units on a scale | -5.4 (1.21) | -6.2 (1.12)

2. Secondary Outcome: Mean Change From Baseline in 10-Item Version of Neuropsychiatric Inventory (NPI-10) at Week 12
Description: NPI assessed noncognitive psychopathology in participants with Alzheimer's dementia. A 10-item scale of the standard 12-item NPI measured neuropsychiatric symptoms minus the appetite and sleep disturbance items. Scores for each subscale (frequency × severity) were calculated to obtain the item score. The total subscale score ranged from 0 to 120, with higher scores indicating more frequent and/or severe A/A symptoms. If a symptom was not present at all, the site would not enter anything for frequency or severity, and a zero would be imputed for that item. LS Mean value was adjusted for NPI strata, treatment, pooled site, visit, treatment-by-visit, baseline NPI-10, and baseline-by-visit interaction.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY451395 | Placebo
Number analyzed (Participants) | 43 | 50
units on a scale | -8.2 (2.08) | -9.3 (1.93)

3. Secondary Outcome: Mean Change From Baseline in the Neuropsychiatric Inventory (NPI) Depression Domain at Week 12
Description: NPI Depression domain was an item of the standard 12-item NPI that measured depression in participants with Alzheimer's dementia. Scores for each subscale (frequency × severity) were calculated to obtain the item score, which ranged from 0 to 12 with higher scores indicating more frequent and/or severe neuropsychiatric symptoms. If a symptom was not present at all, the site would not enter anything for frequency or severity, and a zero would be imputed for that item. LS Mean value was adjusted for NPI strata, treatment, pooled site, visit, treatment-by-visit, baseline NPI depression, and baseline-by-visit interaction.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY451395 | Placebo
Number analyzed (Participants) | 43 | 50
units on a scale | -0.2 (0.34) | -1.0 (0.32)

4. Secondary Outcome: Mean Change From Baseline in the Neuropsychiatric Inventory (NPI) Psychosis Subscale Score at Week 12
Description: The NPI Psychosis subscale score was the sum of the delusions and hallucinations items of the standard 12-item NPI that measured psychosis symptoms in participants with Alzheimer's dementia. Scores for each subscale (frequency x severity) were calculated for each item score and ranged from 0 to 24 with higher scores indicating more frequent and/or severe neuropsychiatric symptoms. LS Mean value was adjusted for NPI strata, treatment, pooled site, visit, treatment-by-visit, baseline NPI psychosis, and baseline-by-visit interaction.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY451395 | Placebo
Number analyzed (Participants) | 43 | 50
units on a scale | -0.4 (0.58) | -0.4 (0.54)

5. Secondary Outcome: Mean Change From Baseline in Cohen-Mansfield Agitation Inventory-Community Version (CMAI-C) at Week 12
Description: CMAI-C is the Cohen-Mansfield Agitation Inventory - Community Version, and it contained 36 questions. The first 35 items were rated from 1 (never) to 7 (several times per hour) and the last item asked if there was any other inappropriate behavior, with a free text field to specify the behavior. The total score ranged from 7 to 245 (7 x 35), with higher scores reflecting more severe agitation. LS Mean value was adjusted for NPI strata, treatment, pooled site, visit, treatment-by-visit, baseline CMAI-C, and baseline-by-visit interaction.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY451395 | Placebo
Number analyzed (Participants) | 42 | 50
units on a scale | -7.2 (1.98) | -4.1 (1.79)

6. Secondary Outcome: Mean Change From Baseline in Cornell Scale for Depression in Dementia (CSDD) at Week 12
Description: CSDD was a 19-item, clinician-rated scale designed to measure the presence and severity of depressive symptoms in dementia participants. Symptoms were rated as absent, mild/intermittent, or severe. Scores ranged from 0 to 38; scores of 8 or more suggested clinical depression. LS Mean value was adjusted for NPI strata, treatment, pooled site, visit, treatment-by-visit, baseline CSDD, and baseline-by-visit interaction.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY451395 | Placebo
Number analyzed (Participants) | 39 | 47
units on a scale | -2.5 (0.59) | -2.7 (0.54)

7. Secondary Outcome: Mean Change From Baseline in Total T-Score in the Frontal System Behaviors Scale (FrSBe) at Week 12
Description: FrSBe was a 46-item, caregiver-rated scale that assessed behaviors associated with damage to the frontal lobes and frontal systems of the brain, including executive function, disinhibition, and apathy. Raw scores were normalized to T-scores based on gender, education, and age. Higher T scores represent a worse outcome. A score of 50 reflects a normative sample, and T scores at or above 65 are considered clinically significant. LS Mean value was adjusted for NPI strata, treatment, pooled site, visit, treatment-by-visit, baseline FrSBe, and baseline-by-visit interaction.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY451395 | Placebo
Number analyzed (Participants) | 42 | 49
units on a scale | -2.2 (2.02) | 2.3 (1.88)

8. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression-Severity-Agitation/Aggression (CGI-S-A/A) at Week 12
Description: CGI-S-A/A was a 7-point, single-item rating scale for overall severity of symptoms based on the investigator's general clinical experience with a similar participant population. This Likert scale ranged from 0 (normal) to 7 (most severely ill). LS Mean value was adjusted for NPI strata, treatment, pooled site, visit, treatment-by-visit, baseline CGI-S-A/A, and baseline-by-visit interaction.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY451395 | Placebo
Number analyzed (Participants) | 43 | 50
units on a scale | -0.7 (0.15) | -0.6 (0.14)

9. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression-Severity-Global Functioning (CGI-S-GF) at Week 12
Description: CGI-S-GF was a 7-point, single-item rating scale for overall functioning based on the investigator's general clinical experience with a similar participant population. This Likert scale ranged from 0 (normal) to 7 (most severely ill). LS Mean value was adjusted for NPI strata, treatment, pooled site, visit, treatment-by-visit, baseline CGI-S-GF, and baseline-by-visit interaction.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY451395 | Placebo
Number analyzed (Participants) | 43 | 50
units on a scale | -0.2 (0.11) | -0.03 (0.11)

10. Secondary Outcome: Mean Change From Baseline in the 14-Item Alzheimer's Disease Assessment Scale, Cognitive Subscale (ADAS-Cog14) at Week 12
Description: ADAS-Cog14, a 14-item rating scale, measured the severity of cognitive dysfunction in persons with AD. Scores ranged from 0 to 90, with a higher score indicating worse cognitive functioning. LS Mean value was adjusted for NPI strata, treatment, pooled site, visit, treatment-by-visit, baseline ADAS-Cog, and baseline-by-visit interaction.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY451395 | Placebo
Number analyzed (Participants) | 43 | 49
units on a scale | -0.1 (0.98) | -0.6 (0.92)

ADVERSE EVENTS:
Groups:
- LY451395 Acute Treatment: 3 milligram (mg) LY451395 orally twice daily for 12 weeks; may have been reduced to 1 mg if participant was unable to tolerate.
- Placebo Acute Treatment: Placebo orally twice daily for 12 weeks
- LY451395 Washout: A 1-week single-blind washout period after the acute period, during which time all randomized participants received placebo.
- Placebo Washout: A 1-week single-blind washout period after the acute period, during time which all randomized participants received placebo.
- LY451395 Post-Study; Placebo Post-Study: The 30-day period after a participant had taken the last dose of study drug, during which time serious adverse event (SAE) information was collected.
Arm/Group | LY451395 Acute Treatment | Placebo Acute Treatment | LY451395 Washout | Placebo Washout | LY451395 Post-Study | Placebo Post-Study
Serious Adverse Events (participants affected / at risk) | 5/63 | 4/69 | 0/42 | 0/49 | 1/63 | 0/69
Other Adverse Events (participants affected / at risk) | 24/63 | 24/69 | 1/42 | 2/49 | 0/63 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY451395 Acute Treatment (N=63) | Placebo Acute Treatment (N=69) | LY451395 Washout (N=42) | Placebo Washout (N=49) | LY451395 Post-Study (N=63) | Placebo Post-Study (N=69)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY451395 Acute Treatment (N=63) | Placebo Acute Treatment (N=69) | LY451395 Washout (N=42) | Placebo Washout (N=49) | LY451395 Post-Study (N=63) | Placebo Post-Study (N=69)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1/31 (1) | 0/36 (0) | 0/22 (0) | 0/27 (0) | 0/31 (0) | 0/36 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0/32 (0) | 1/33 (1) | 0/20 (0) | 0/22 (0) | 0/32 (0) | 0/33 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days